CLINICAL TRIAL: NCT06673277
Title: Skin Temperature Response to Prolonged Cooling With an Electronic Continuous Cold-flow Cryocompression Device: a Safety and Feasibility Pilot
Brief Title: Prolonged Cryocompression and Skin Temperature: a Safety and Feasibility Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Winchester (Other)
Collaborators: Physiolab Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HWB_REC_2405_Belsey
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Skin Temperature Change; Adverse Effects; Safety of Intervention; Cryotherapy; Feasibility Pilot Study
Keywords: skin temperature; cryotherapy; cryocompression; safety; feasibility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prolonged cooling at 8 ℃ then 10 ℃ (Experimental): The device will be set to circulate water through the cuff around the knee at 8 ℃ for the first 30-minutes, then at 10 ℃ for the subsequent 90-minutes.
  Interventions: Device: Prolonged (2-hour) cryocompression therapy
- Prolonged cooling at 8 ℃ then 12 ℃ (Experimental): The device will be set to circulate water through the cuff around the knee at 8 ℃ for the first 30-minutes, then at 12 ℃ for the subsequent 90-minutes.

INTERVENTIONS:
Device: Prolonged (2-hour) cryocompression therapy — The cuff of the device will be attached around the knee randomised to receive the treatment as per the manufacturer's instruction. Then the device will be set to apply a standard 30-minute treatment with a temperature of 8 ℃ and intermittent compression of 25-50 mmHg. Following this, and depending on the randomised condition, the treatment will continue for a further 90-minutes with a temperature of either 10 ℃ or 12 ℃ being applied by the device. The level of compression will remain the same (25-50 mmHg) throughout all tests.
  Arms: Prolonged cooling at 8 ℃ then 10 ℃

SUMMARY:
Guidelines for treatment duration for cold and compression therapy after knee surgery are typically based on the use of ice packs for 30 minutes. However, electronic devices are beginning to be used more commonly in post-operative settings and while they have been shown to be able to provide a therapeutic dose of cooling, the necessary reduction in tissue temperature to realise the benefits of the therapy is much more gradual than ice packs and takes a longer time. Therefore, longer treatment durations may be needed with electronic devices. Although other research has demonstrated that skin temperature can be safely cooled continuously for several hours, no study has done this with an electronic device and monitored whether skin temperature is controlled to remain with a known therapeutic range of 10-15 ℃.

This pilot study aims to test the feasibility and safety of a 2-hour treatment duration while skin temperature around the knee of 15-17 healthy volunteers is recorded. Each participant will take part in two treatments, whereby the first 30-minutes of both treatments involves cooling at a temperature of 8 ℃ (known to effectively reduce skin temperature), immediately followed by 90 minutes of cooling at either 10 ℃ or 12 ℃ (depending on the treatment condition) with the aim of maintaining skin temperature within the 10-15 ℃ target range. At least 24 hours will be left in between treatments with same participant.

DETAILED DESCRIPTION:
Introduction Despite the advancement in technology for cryocompression therapy in rehabilitation after knee surgery, guide-lines for the duration of cryocompression treatments, remain largely unchanged at typically 15-30 minutes in length (Long and Jutte, 2020). This duration was originally established with the traditional use of ice packs, which provide rapid cooling and must be limited to this relatively short time period to reduce the likelihood of cold-related complications or injury (MacAuley, 2001; Wilke and Weiner, 2003; Thienpont, 2014). Electronic devices have been shown to reduce tissue temperature more gradually, and to provide an effective dose of cold without lowering tissue temperature to potentially unsafe levels (Belsey, Reid, et al., 2024). Consequently, the traditional treatment duration guidelines may not be relevant for electronic devices.

Prolonged cooling durations are more likely to effect pain and inflammation around deeper tissues (Long and Jutte, 2020), which could lead to improvements in post-operative clinical outcomes. Exposure to cold of 15 ℃ using a non-electronic technology for up to 6 hours has previously been demonstrated as safe (Kwiecien, McHugh and Howatson, 2020). One study investigated prolonged cooling (3 hours per treatment) with an elec-tronic device following knee surgery and although no complications were reported, skin temperature response was not measured. Therefore, despite safety being indicated, it is not known whether an optimal dose of cooling was applied that reduced skin temperature to within an established optimal therapeutic zone of 10-15 ℃ (Wilke and Weiner, 2003; Bleakley and Hopkins, 2010).

The safety and feasibility of prolonged exposure to cryocompression with an electronic device that is known to provide an effective dose of cold has not explicitly been examined, and should be established if traditional treat-ment duration guidelines are to be challenged, amended, and optimised for this therapy modality. Therefore, the aim of this study is to investigate the ability of an electronic cryocompression device to maintain skin tempera-ture within the target therapeutic zone for a prolonged period, and to assess the safety and feasibility of such a treatment protocol. The results from this exploratory pilot study can then be used for future research into the efficacy of prolonged cooling in clinical settings and investigations into optimal treatment duration depending on the therapy modality employed.

It is hypothesised that an electronic cryocompression device will successfully reduce skin temperature will be re-duced and maintained within the 10-15 ℃ target range during a prolonged treatment. Secondly, it is predicted that there will be no treatment-related adverse events and the protocol will be well tolerated by participants in terms of perceived comfort.

Methods Design This prospective randomised controlled crossover trial will recruit healthy adult volunteers from a university population to participate, in line with previously published recommendations for appropriate sample sizes for pilot studies (Julious, 2005; Johanson and Brooks, 2010). Each participant will take part in each of the two conditions in order to eliminate the risk of demographic factors confounding the results. Conditions will be conducted in a random order, as determined by a random number generator before recruitment begins. Conditions will involve the application of a Physiolab S1 cryocompression device in accordance with the manufacturers' guidelines. Each testing session will take around 3 hours to complete, with at least 24 hours between tests with the same participant. In total, participants will be giving no more than 6 hours of time across 2 days to complete their participation. Participants will not be compensated for taking part in the study, nor will they be charged.

Protocol All eligible participants will first be required to provide informed consent prior to their participation in the study, and will be asked to avoid caffeine, tobacco, and strenuous exercise within the 2 hours prior to testing. The height and mass of the participants will be measured at the beginning of the first test session in order to calculate BMI, and participants' age and sex will be recorded to allow for later analysis to determine any confounding influence of these factors on the results.

Participants will then be asked to lie supine on a physiotherapy bed for 20-minutes to allow body temperature to acclimatise to the test environment and to ensure that the feet are at the same level as the heart, which is important for the capillary refill test that will be conducted on the second toe of the leg that receives cryotherapy, multiple times throughout the study period. During the 20-minute acclimatisation period, the following anatomical landmarks on the treatment leg will be marked with a small square of micropore tape in preparation for the range-of-motion measurements that will be taken before and after the cryotherapy treatment: greater trochanter, lateral epicondyle, and lateral malleolus. Additionally, the acclimatisation period will also be used to prepare and affix 3 iButton temperature sensors to the treatment leg with more micropore tape: one 20 mm distal to the patella, one in an equivalent position posteriorly, and one on the plantar side of the proximal pulp of the big toe. The two iButtons positioned about the knee have been shown to have the highest reproducibility for human skin temperature measurement around that joint (Priego-Quesada et al., 2021) and will measure changes directly within the cryocompression treatment area. Measurements taken by the iButton on the toe will be used in combination with the results of the capillary refill tests to monitor changes in perfusion as a safety measure during prolonged cryocompression, and to ensure a return to normal following the treatment. The iButton is a small temperature sensor that has been validated for human skin temperature measurement (van Marken Lichtenbelt et al., 2006; Smith et al., 2010). The leg that will be used for the study will be randomly selected for each participant, and will remain the same for each condition.

Following the acclimatisation period, a capillary refill test will be conducted on the second toe and skin temperature of the big toe will be measured. A measurement of range-of-motion from extension to flexion will also be taken at this time using a standard goniometer. These measures taken prior to the cryocompression treatment will provide the reference baseline values that will be monitored to ensure the safety of the participant and to detect any abnormal response to the prolonged cooling protocol. Baseline skin temperature measurements around the knee will also be recorded at this point.

Once the baseline measures have been taken, the cryocompression device will then be applied to the leg of the participant and the treatment will begin. The first 30 minutes of each test will involve the device being set to circulate cold water at 8 ℃, as this has been shown to reduce skin temperature to within the target 10-15 ℃ range with this device (Belsey, Gregory, et al., 2024). The device will continue to provide a treatment for an additional 90 minutes with water temperature adjusted to either 10 ℃ or 12 ℃, depending on the randomised condition being tested. These temperatures have been chosen to reflect the minimum and maximum temperatures that the device is able to apply that fall within the target skin temperature range. Choosing a water temperature <10 ℃ for prolonged cooling would risk skin temperature dropping to below the target range, as equilibrium may be approached, which could increase the risk of adverse events (Wilke and Weiner, 2003). The device will apply intermittent compression of 25-50 mmHg consistently throughout each test, in line with the manufacturer-recommended setting for knee treatments.

Every 30 minutes, the cuff of the device will briefly be removed from the leg of the participant to inspect the skin for any indication of an abnormal reaction. To compliment this visual inspection, a pain rating will be concurrently recorded using a Numerical Pain Rating Scale (NPRS), along with another capillary refill test and skin temperature measurement of the toe. If any adverse events are identified or suspected based on the visual inspection, or if pain scores exceed 5/10 at any time, or if the capillary refill test lasts longer than 6 seconds for two consecutive measurements during the treatment period, the test will be terminated and the participant will take no further part in the study. In addition to the safety checks, a perceived rating of comfort will simultaneously be recorded every 30 minutes by responding to the following question using a 5-point Likert scale: "How would you rate the comfort of the treatment?" The possible answers to this question will be: "Very comfortable, Comfortable, Neutral, Uncomfortable, Very uncomfortable". This will provide insight into differences in tolerance of the treatment, which could be relevant for the feasibility of a prolonged cooling protocol in clinical settings.

Following the 2-hour prolonged cooling treatment, the cuff will be removed from the participant and skin temperature will continue to be measured every 5 minutes for a further 15 minutes, as this is the maximum length of time it is expected that skin temperature will remain <15 ℃ while the leg re-warms (Belsey, Gregory, et al., 2024). This will allow for the total time to be measured that skin temperature remains within the target therapeutic range as a result of the cryocompression treatment. At the point of cuff removal and 15 minutes lat-er, capillary refill tests will once again be conducted to monitor the expected normalisation of perfusion of the treatment leg. Normalisation will be defined by capillary refill times are less than 3 seconds in participants under 50 years, and less than 4.5 seconds in participants over 50 years to account for normal age-related differ-ences. 15 minutes after the treatment, a second range-of-motion test will be performed in the same fashion as before to determine whether there is any residual stiffness/weakness as a result of the treatment. Functionally meaningful changes in range-of-motion of the knee have been suggested to be >5 °, so a return to "normal" range-of-motion will be established if the post-test score is within 5 ° of the baseline measure. At this point, a final pain and comfort rating will be recorded and the temperature sensors will be removed from the leg of the participant; thus ending their participation in the test. If the results of the capillary refill test or range-of-motion measurement have not returned to normal as defined above, the treatment leg will be actively re-warmed by being placed in a water bath at 38 ℃ for a further 15 minutes. The capillary refill test and range-of-motion will be measured again at the end of this subsequent 15-minute period. If results have still not returned to within normal parameters, and the participant or researcher has concerns, then medical advice will be sought and attention provided as necessary. Otherwise, the participant will be allowed to leave the lab but will be contacted by the researcher two hours later (by a contact method chosen by the participant) to enquire as to whether there have been any changes. At which point, medical advice can be recommended or sought, if needed. Once each participant has taken part in all conditions, they will have completed their participation in the study .

Analysis The data will be analysed to detect any differences during testing compared to baseline measures, and between groups. All data will be first subjected to a Kolmogorov-Smirnov test to assess whether they are normally distributed. A repeated measures analysis of variance will be performed on all normally distributed data. A Friedman test will be performed on any data that are not normally distributed .

Ethical issues Although this is a safety study and adverse events will be monitored as outcomes, the risk of any being identified is deemed to be low. Individuals will be screened prior to participation to ensure that nobody who would otherwise be contraindicated for cryocompression therapy is recruited. The temperature settings used during treatments were chosen as they are expected to reduce and maintain skin temperature within the target zone, while preventing it from dropping below the 10 ℃ threshold where the risk of complications is increased. Additionally, a previous study reported no cold-related complications when skin temperature was maintained at 7 ℃ continuously for 2 hours (Morsi, 2002), suggesting that the 10 ℃ threshold is cautious. Similarly, a 2-hour treatment duration has been chosen as a conservative time period for prolonged cooling, as other methods have been safely applied for much longer durations, as outlined in the introduction. Nevertheless, this will be the first time an electronic device providing a known effective dose of cold for a prolonged period of time has been investigated. Therefore, the temperature settings and treatment duration were chosen to keep risk to the participants at an absolute minimum.

Participants have the right to withdraw themselves and any collected data from the study at any time during participation, and for 7 days after the final test session, without having to give a reason. They also have the right to terminate a test session at any time. After 7 days have passed since a participant's final test session, their data will be anonymised and used as part of the final dataset for analysis. Testing shall also be terminated as a result of any adverse reactions that emerge. Any adverse reactions that occur shall be addressed and monitored, as appropriate, until things return to baseline/normal. If a test is terminated for a reason that could be mitigated in future, participants will be offered the opportunity to repeat the test another day, should they wish to continue taking part in the study. If a test is terminated due to an adverse reaction that can not be mitigated in future, the participant (and any collected data) will be thanked for their time and withdrawn from the study. All members of the research team have been trained to be able to competently use the cryocompression device and to correctly execute the test protocol outlined above. A qualified first aider will always be present within the labs while tests are being conducted, and all lab rules and safety protocols will be followed at all times (e.g. cleaning up water spills).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years

Exclusion Criteria:

* BMI >40 kg/m2
* History of nerve damage or sensory deficit in the lower limbs (including frostbite)
* Hypersensitivity to cold, including hives
* Active inflammation or pain of the knee
* History of thrombosis, embolism, or other conditions related to impaired peripheral circulation
* Suffering from diagnosed diabetes, multiple sclerosis, rheumatoid arthritis, spinal cord injury, cardio-vascular disease, hypertension, Raynaud disease, cryoglobulinemia, or haemoglobinuria
* Confirmed or suspected tissue infection, an unstable fracture, a skin condition, or a tumour in the treatment area
* Cognitive impairment or communication barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Skin temperature of the knee | From the baseline measurement immediately prior to the treatment, then every 5 mins during the treatments, until a maximum of 30 minutes following the end of the treatment. This timeframe will apply to both treatments that participants will receive.
  Measured in ℃ using 2 iButton temperature sensors attached with microporous tape. One positioned 20 mm distal to the patella, and one positioned in an equivalent location on the back of the leg.

SECONDARY OUTCOMES:
Skin temperature of the toe | From the baseline measurement immediately prior to the treatment, then every 30 mins during the treatments, then at 15 and 30 minutes following the end of the treatment. This timeframe will apply to both treatments that participants will receive.
  Measured in ℃ on the underside of the big toe on the treatment leg. This is part of the safety monitoring in combination with the capillary refill tests that will help to establish that normal blood flow has returned through the treatment leg following each test.
Normalisation of perfusion of the toe | Once at baseline immediately prior to the test, then every 30 minutes during each test, and at 15 and 30 minutes following each test.
  A capillary refill test will be performed on the second toe of the treatment leg as part of the safety monitoring to ensure a return to normal blood flow of the treatment leg following each test. If refill time takes >6 seconds for 2 consecutive tests, then the treatment will be terminated.
Range-of-motion of the knee | Once at baseline immediately prior to the test, then 15 and 30 minutes following the treatment. This will be repeated for each of the 2 tests participants receive.
  Measured with a goniometer as part of the safety monitoring to ensure a return to normal function following each test.
Perceived pain | At baseline immediately prior to the test, then every 30 minutes during the treatment, and after 15 and 30 minutes following each treatment.
  Using a Numerical Pain Rating Scale where 0 equals "no pain" and 10 equals "the most severe pain possible", participants will report any pain sensations they experience during testing. This is part of the safety monitoring process and a test will be terminated if pain scores reach 5/10 or greater. Participants will be blinded to this threshold for test termination.
Adverse effects | At baseline immediately prior to testing, then every 30 minutes during treatments, and after 15 and 30 minutes following treatments.
  A visual inspection of the leg periodically throughout each test will be conducted to monitor any unexpected adverse effects that may occur in response to the treatment (e.g. unusual discolouration of the treatment area). Tests will be terminated upon the occurrence of any of these type of adverse effects. None are expected due to the exclusion criteria of the study ensuring that individuals who would be contraindicated for cryocompression, due to relevant risk factors, do not take part.
Perceived comfort | Every 30 minutes during a treatment, and after 15 and 30 minutes following each test.
  Ratings of comfort will be provided by choosing 1 of 5 potential answers to the following question "How would you rate the comfort of the treatment?". The possible answers are: "Very comfortable, Comfortable, Neutral, Uncomfortable, Very uncomfortable".

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hannah, PhD, Principal Investigator — University of Winchester
Locations (1):
- University of Winchester, Winchester, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All individual participant data will remain within the study site and only accessible by the research team. Upon completion of the study, all data will be anonymised and aggregated for analysis. It is the results of the analyses - providing information relating to group averages - that will be shared within a manuscript that is eventually published in a peer-reviewed journal, or mentioned within professional conference presentations.

REFERENCES:
- [Background] Wilke B, Weiner RD. Postoperative cryotherapy: risks versus benefits of continuous-flow cryotherapy units. Clin Podiatr Med Surg. 2003 Apr;20(2):307-22. doi: 10.1016/S0891-8422(03)00009-0. PMID 12776983
- [Background] Waterman B, Walker JJ, Swaims C, Shortt M, Todd MS, Machen SM, Owens BD. The efficacy of combined cryotherapy and compression compared with cryotherapy alone following anterior cruciate ligament reconstruction. J Knee Surg. 2012 May;25(2):155-60. doi: 10.1055/s-0031-1299650. PMID 22928433
- [Background] Thienpont E. Does advanced cryotherapy reduce pain and narcotic consumption after knee arthroplasty? Clin Orthop Relat Res. 2014 Nov;472(11):3417-23. doi: 10.1007/s11999-014-3810-8. Epub 2014 Jul 25. PMID 25059851
- [Background] Smith AD, Crabtree DR, Bilzon JL, Walsh NP. The validity of wireless iButtons and thermistors for human skin temperature measurement. Physiol Meas. 2010 Jan;31(1):95-114. doi: 10.1088/0967-3334/31/1/007. Epub 2009 Nov 26. PMID 19940348
- [Background] Selfe, J. et al. (2009) 'An investigation into the effect on skin surface temperature of three cryotherapy modali-ties', Thermology International, 19(4), pp. 119-124.
- [Background] Priego-Quesada JI, Gandia-Soriano A, Pellicer-Chenoll MT, Catala-Vilaplana I, Bermejo-Ruiz JL, Encarnacion-Martinez A, Salvador-Palmer R, Cibrian Ortiz de Anda R. Reproducibility of Skin Temperature Response after Cold Stress Test Using the Game Ready System: Preliminary Study. Int J Environ Res Public Health. 2021 Aug 5;18(16):8295. doi: 10.3390/ijerph18168295. PMID 34444044
- [Background] Morsi E. Continuous-flow cold therapy after total knee arthroplasty. J Arthroplasty. 2002 Sep;17(6):718-22. doi: 10.1054/arth.2002.33562. PMID 12216025
- [Background] van Marken Lichtenbelt WD, Daanen HA, Wouters L, Fronczek R, Raymann RJ, Severens NM, Van Someren EJ. Evaluation of wireless determination of skin temperature using iButtons. Physiol Behav. 2006 Jul 30;88(4-5):489-97. doi: 10.1016/j.physbeh.2006.04.026. Epub 2006 Jun 23. PMID 16797616
- [Background] Mac Auley DC. Ice therapy: how good is the evidence? Int J Sports Med. 2001 Jul;22(5):379-84. doi: 10.1055/s-2001-15656. PMID 11510876
- [Background] Long, B.C. and Jutte, L.S. (2020) '21st Century Attacks on Cryotherapy in Sports Health Care-Clinician Be-ware', Athletic Training & Sports Health Care, 12(3), pp. 99-101. Available at: https://doi.org/10.3928/19425864-20200401-02.
- [Background] Kwiecien SY, McHugh MP, Howatson G. Don't Lose Your Cool With Cryotherapy: The Application of Phase Change Material for Prolonged Cooling in Athletic Recovery and Beyond. Front Sports Act Living. 2020 Oct 15;2:118. doi: 10.3389/fspor.2020.00118. eCollection 2020. PMID 33345107
- [Background] Julious, S.A. (2005) 'Sample size of 12 per group rule of thumb for a pilot study', Pharmaceutical Statistics, 4(4), pp. 287-291. Available at: https://doi.org/10.1002/pst.185.
- [Background] Johanson, G.A. and Brooks, G.P. (2010) 'Initial scale development: Sample size for pilot studies', Educational and Psychological Measurement, 70(3), pp. 394-400. Available at: https://doi.org/10.1177/0013164409355692.
- [Background] Fang L, Hung CH, Wu SL, Fang SH, Stocker J. The effects of cryotherapy in relieving postarthroscopy pain. J Clin Nurs. 2012 Mar;21(5-6):636-43. doi: 10.1111/j.1365-2702.2010.03531.x. Epub 2011 Feb 20. PMID 21332855
- [Background] Bleakley, C.M. and Hopkins, J.T. (2010) 'Is it possible to achieve optimal levels of tissue cooling in cryothera-py?', Physical Therapy Reviews, 15(4), pp. 344-350. Available at: https://doi.org/10.1179/174328810X12786297204873.
- [Background] Belsey J, Gregory R, Paine E, Faulkner J. Skin temperature of the knee was effectively reduced when using a new continuous cold-flow cryocompression device: a randomised controlled crossover trial. Physiotherapy. 2024 Jun;123:11-18. doi: 10.1016/j.physio.2023.12.001. Epub 2023 Dec 14. PMID 38244486
- [Background] Belsey J, Reid A, Paine E, Faulkner J. A randomised crossover trial of five cryocompression devices' ability to reduce skin temperature of the knee. PLoS One. 2024 Jan 16;19(1):e0296634. doi: 10.1371/journal.pone.0296634. eCollection 2024. PMID 38227605